CLINICAL TRIAL: NCT04152122
Title: A Novel Dynamic Random-dot Stereopsis Assessment to Measure the Stereopsis in Intermittent Exotropia
Status: Completed | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Clinical Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2016MEKY032
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Dynamic Stereopsis in Intermittent Exotropia Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intermittent exotropia group: Intermittent exotropia group
  Interventions: Diagnostic Test: The dynamic stereopsis test
- Normal group: Normal group
  Interventions: Diagnostic Test: The dynamic stereopsis test

INTERVENTIONS:
Diagnostic Test: The dynamic stereopsis test — The characteristics of preoperative dynamic stereopsis in 83 intermittent exotropia patients and its associations with clinical features were analysed, and the prognosis was followed up on the 1st day and 2nd, 6th and 12nd months postoperatively.

SUMMARY:
A novel dynamic random-dot stereopsis test that included motion + disparity (MD), motion (M), and disparity (D), in which the disparity cues range from 200 to 1200 arc-seconds was used. The characteristics of preoperative dynamic stereopsis in 83 intermittent exotropia patients and its associations with clinical features were analysed, and the prognosis was followed up on the 1st day and 2nd, 6th and 12nd months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

X(T) groups were as follows:

1. near and distance exodeviation angles greater than 5 prism degrees (PD) and alternate cover tests and X(T) diagnosis by an experienced doctor;
2. between 5 and 30 years old;
3. 0.0 or better best corrected visual acuity (BCVA; logMAR, log of the minimum angle of resolution);
4. absence of other ocular disorders or other systemic diseases.

Normal group were as follows:

1. between 5 and 30 years old;
2. 0.0 or better logMAR BCVA;
3. near and distance exodeviation angles less than 5 PD and alternate cover tests; and
4. no history of any ocular pathology or systemic disease.

Exclusion Criteria:

X(T) groups were as follows:

1. near and distance exodeviation angles less than 5 prism degrees (PD)
2. younger than 5 or older than 30 years old;
3. less than 0.0 or better best corrected visual acuity (BCVA; logMAR, log of the minimum angle of resolution);
4. has other ocular disorders or other systemic diseases.

Normal group were as follows:

1. younger than 5 or older than 30 years old;
2. less than 0.0 or better best corrected visual acuity (BCVA; logMAR, log of the minimum angle of resolution);
3. near and distance exodeviation angles more than 5 PD and alternate cover tests;
4. has history of any ocular pathology or systemic disease.

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A total of 83 cases X(T) patients and 50 normal subjects were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
The mean reciprocal value of stereopsis | 1st day
  The mean reciprocal value of stereopsis on the 1st day
The mean reciprocal value of stereopsis | 2nd month
  The mean reciprocal value of stereopsis on the 2nd month
The mean reciprocal value of stereopsis | 6th month
  The mean reciprocal value of stereopsis on the 6th month
The mean reciprocal value of stereopsis | 12th month
  The mean reciprocal value of stereopsis on the 6th month

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Opthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
A novel dynamic random-dot stereopsis test that included motion + disparity (MD), motion (M), and disparity (D), in which the disparity cues range from 200 to 1200 arc-seconds was used. The characteristics of preoperative dynamic stereopsis in 83 intermittent exotropia patients and its associations with clinical features were analysed, and the prognosis was followed up on the 1st day and 2nd, 6th and 12nd months postoperatively.